CLINICAL TRIAL: NCT01753427
Title: Perception of Symptom Variability in Chinese COPD Patients
Brief Title: Perception of Symptom Variability in COPD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RCN-XXX-2012/1
Record Dates: First submitted 2012-12-13; First posted 2012-12-20 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD,; symptoms,; Non-Interventional study,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The objective of the study is to assess patient's perception with stable state COPD on symptom variability and to describe how symptom variability impacts daily quality of life in Chinese COPD patient with moderate, severe or very severe airflow limitation from tier 3 hospitals in China where most of COPD patients are diagnosed and treated.

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent
* Out-patient
* Clinical diagnosis of COPD at least 6 months
* Lung function based on data available within 3 months in medical records confirming FEV1<80% normal predicted (post-bronchodilator) and FEV1/FVC<0.7 (post-bronchodilator)

Exclusion Criteria:

* Participation in any interventional study involving investigational drugs; Patient inability to understand the study procedures or inability/reluctance to answer questionnaire
* Ongoing exacerbation of COPD or exacerbation within the previous 3 months. An exacerbation is defined as a worsening of COPD symptoms leading to a treatment with antibiotics and/or a short course of system steroids and/or hospitalisation or emergency
* History of asthma and/or allergic rhinitis, Lung cancer or any other significant respiratory disease such as bronchiectasis, lung fibrosis, interstitial lung disease, tuberculosis, sarcoidosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out-patient, male or female aged 40 years and over and Clinical diagnosis of COPD at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 1058 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The variability of symptoms due to COPD throughout the day | Day 1
  * To ask subject, which symptoms（breathlessness, chest tightness, coughing, wheezing, phlegm）is COPD symptoms and exist throughout the day
  * To ask subject , whether COPD symptoms variability throughout the day exists or not ;
  * To ask subject , which (on waking, later in the morning, in the afternoon, in the evening, at night) is the most likely occurring time of these symptoms;
  * To ask subject , Which (on waking, later in the morning, in the afternoon, in the evening, at night) is the most troublesome time of these symptoms.

SECONDARY OUTCOMES:
The impact of COPD symptoms on patient's daily living activities and sleep quality | Day 1
  * To ask subject, Whether essential daily activities affected by COPD symptoms and the type of following: going up and downstairs, Going out of shopping, doing sport/exercise, doing housework, or all of these
  * To ask subject, Whether sleep quality affected by COPD symptoms and the type of following: difficulty falling sleep, frequent waking during night, early waking in the morning, or all of these
The impact of COPD symptoms on morning activities | Day 1
  * To ask subject, When [getting out of bed, dressing, washing, eating breakfast, morning activity after breakfast (indoor activity, including housework) , morning exercise (outdoor activity, such as walking, sport, etc)] the essential morning activities affected by COPD symptoms:
  * To ask subject, The extent of these morning activities affected: not at all, a little, moderate, severe, extremely severe resulting to feel difficult to complete independently, extremely severe resulting to complete under others help or cannot complete at all
Total CAT score | Day 1
  CAT (COPD assessment test) has a broader coverage of the impact of COPD on the patient's daily life and well-being.
Total MMRC score | Day 1
  MMRC (Modified Medical Research Council Questionnaire for Assessing the Severity of Breathlessness) assesses disability due to breathlessness.
Patient's perception on COPD and COPD treatments | Day 1
  * To ask subject, Seek for treatment only when symptoms occur/worsening or regularly visit physician and take medicine(s)
  * To ask subject, Whether Knowing about how and when to use their medications
  * To ask subject, Usually taking their medication(s) required by physician to be used in the morning at what time: before getting out of bed, within 30 minutes after getting out of bed, within 30 minutes to 1 hour after getting out of bed, over 1 hour after getting out of bed, no regular time

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Wuhan, Hubei
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1036&filename=NIS-RCN-XXX-2012-1_Report_Synopsis.pdf
- See also: YAO Wanzhen et al COPD symptom NIS abstract_2014 APSR. Abstract ID: P-F-090 — http://onlinelibrary.wiley.com/doi/10.1111/resp.12417_6/epdf